CLINICAL TRIAL: NCT00192608
Title: A 48-Week, Randomised, Study to Describe the Pharmacokinetic Profile and Durability of Atazanavir-Saquinavir-Ritonavir Once Daily and Describe the Pharmacokinetic Profile of Saquinavir-Ritonavir Using Saquinavir 500mg Formulation.
Brief Title: A 48-Week, Randomised, Study to Describe the Pharmacokinetic Profile and Durability of Atazanavir-Saquinavir-Ritonavir Once Daily and Describe the Pharmacokinetic Profile of Saquinavir-Ritonavir Using Saquinavir 500mg Formulation: the ASK-500 Study
Acronym: ASK-500
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: The University of New South Wales, University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASK-500 14047; ACTR012605000660684
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: HIV Infections
Keywords: Pharmacokinetics, atazanavir, saquinavir, ritonavir, HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- saquinavir at baseline (Experimental): patients receiving NRTIs + saquinavir + ritonavir 1000/100 mg BID at entry switch from 200 mg SQV capsules to 500 mg SQV tablets following PK at day 0. After PK at day 8 NRTIs ceased and regimen changed to ATV/SQV/RTV 300/1500/100 QD using 500 mg SQV formulation and continued to week 48
  Interventions: Drug: saquinavir 500 formulation
- other boosted PI at baseline (Experimental): Patients receiving NRTIs + PI/RTV randomised at baseline to receive ATV/SQVRTV 300/1500/100 QD using 500 mg SQV formulation or ATV/SQV/RTV 300/1600/100 QD using 200 mg formulation. Following PK at day 7, SQV formulation switched with second PK assessment at day 15. Patients then receive ATV/SQV/RTV 300/1500/100 QD to week 48.
  Interventions: Drug: cross-over arm

INTERVENTIONS:
Drug: saquinavir 500 formulation — NRTIs + SQV/RTV 1000/100 mg BID using 200 mg SQV capsules switched at entry to ATV/SQV/RTV 300/1500/100 mg QD using 500 mg SQV tablet for 48 weeks with PK at days 0 and 8.
  Arms: saquinavir at baseline
Drug: cross-over arm — either ATV/SQV/RTV 300/1500/100 QD (500 mg SQV tabs) for 7 days then after PK SQV changed to 1600 mg QD (200 mg caps) with PK day 15, or ATV/SQV/RTV 300/1600/100 QD for 7 days with switch to SQV 1500 mg QD. After day 15 PK both groups switch to ATV/SQV/RTV 300/1500/100 QD to week 48
  Arms: other boosted PI at baseline

SUMMARY:
Saquinavir and Atazanavir are drugs used in combination therapy to treat HIV disease. Saquinavir is currently available in a 200 milligram capsule. Most individuals currently on saquinavir require to take 5 tablets twice a day. In an attempt to reduce this number of pills, a new capsule has been developed containing 500 milligrams of saquinavir. This study will assess: i) blood drug levels in individuals taking both saquinavir formulations, ii) blood drug levels in individuals taking both saquinavir formulations when given with atazanavir, iii) 48 weeks of follow up for individuals receiving the new saquinavir formulation with atazanavir as HIV therapy.

DETAILED DESCRIPTION:
BACKGROUND The development of anti-HIV therapy for the treatment of HIV disease has improved the quality of life and survival of many people with HIV. However the treatments do not always work over long periods, as medications are often difficult to take due to side effects and a large numbers of pills to be taken. This has lead researchers to look for new ways to treat HIV with medications that require fewer numbers of pills and have fewer side effects.

Atazanavir and saquinavir are two drugs used to treat HIV and come from the same class of drugs known as the protease inhibitors. Atazanavir has the advantage of being taken only once a day. Saquinavir is available in a new formulation (type of pill), which will require fewer numbers of pills to be taken daily.

AIM The purpose of this study is to investigate the use of these two drugs used together with ritonavir as a once daily HIV treatment, which will consist of 6 tablets.

Furthermore this study will look at blood drug levels in individuals on atazanavir, saquinavir and ritonavir with and without the new saquinavir formulation to ensure blood levels of these drugs are adequate.

For individuals currently on the old saquinavir formulation, this study will also look at blood drug levels before and after changing to the new formulation.

ELIGIBILITY:
Inclusion Criteria:

HIV-1 infected individuals aged 18 years or over On stable antiretroviral therapy for at least three months consisting of nucleoside reverse transcriptase inhibitors and protease inhibitors OR On stable antiretroviral therapy for at least three months consisting of atazanavir-saquinavir-ritonavir Undetectable HIV RNA viral load for past three months

Exclusion Criteria:

* Individuals receiving on non-nucleoside reverse transcriptase inhibitors within the past three months
* Individuals currently receiving other enzyme inducing agents (as per
* Individuals receiving ritonavir at doses greater than 100 mg bid
* Active AIDS defining illnesses
* Previously documented intolerance or virological failure to saquinavir
* Previously documented intolerance or virological failure to atazanavir
* Patients who are co-infected with Hepatitis B and are likely to require, in their clinician's opinion, HBV nucleoside therapy during the study.
* Female patients who are pregnant, breastfeeding, or who plan to become pregnant during the study
* Any current clinical or laboratory parameter of ACTG Grade 4 (except lipids & CK)
* Evidence of ongoing alcohol and/or drug or substance abuse that would result in the patient being unreliable in fulfilling the conditions of this protocol
* Prior non-adherence to antiretroviral treatment regimens that would result in the patient being unreliable in fulfilling the conditions of this protocol
* Evidence of active opportunistic infection, intercurrent illness, drug toxicity or any other condition that would preclude the patient from taking the prescribed antiretroviral regimen
* Conditions that might interfere with evaluation of the disease under study.
* Conditions/allergies that may compromise the safety of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To compare the pharmacokinectic profile of ATV-SQV-RTV using SQV 500 and 200 formulations. | week 48
To compare the pharmacokinetic profile of SQV/r 1000/100mg bid using SQV 500 and 200 formulations. | week 48
To assess the durability and safety of a once daily double boosted PI regimen comprised of ATV300 - SQV1500 - RTV100 | week 48
To assess the decay pharmacokinetics | week 48

SECONDARY OUTCOMES:
Assessment of adherence to medications. | week 48
Assessment of changes to CD4 lymphocyte count | week 48
Assessment of changes in lipid parameters | week 48
Assessment of changes in monocyte mRNA | week 48

CONTACTS AND LOCATIONS:
Overall Officials: David A Cooper, MD, Principal Investigator — Kirby Institute
Locations (1):
- St Vincents Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Result] Winston A, Mallon PW, Satchell C, MacRae K, Williams KM, Schutz M, Law M, Cooper DA, Emery S. The safety, efficacy, and pharmacokinetic profile of a switch in antiretroviral therapy to saquinavir, ritonavir, and atazanavir alone for 48 weeks and a switch in the saquinavir formulation. Clin Infect Dis. 2007 Jun 1;44(11):1475-83. doi: 10.1086/517507. Epub 2007 Apr 18. PMID 17479946
- See also: National Centre in HIV Epidemiology and Clinical Research Homepage — http://www.med.unsw.edu.au/nchecr/